CLINICAL TRIAL: NCT04735263
Title: Dark Adaptation as an Early Indicator of Response to Statin Therapy for Intermediate AMD
Acronym: DELPHI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, John B. Miller, MD, Assistant Professor of Ophthalmology, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P001265
Record Dates: First submitted 2020-12-23; First posted 2021-02-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: Prospective interventional trial for off label use of FDA approved drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intermediate Age-Related macular degeneration patients (Other): Subjects can have either:
  1. Bilateral high-risk iAMD
  2. High-risk iAMD in one eye with GA and/or CNV in the fellow eye No control arm
  Interventions: Drug: Atorvastatin 80mg

INTERVENTIONS:
Drug: Atorvastatin 80mg — Patient will be receiving 80mg of Atorvastatin, if they are able to tolerate it from the start to the end of the study.
  Other Names: Lipitor 80 mg(Brand name)

SUMMARY:
interventional trial for off label use of high dose atorvastatin 80 mg in intermediate AMD patients and correlate recovery response measured by dark adaptation recovery time with drusen volume reduction measured by SD-OCT

DETAILED DESCRIPTION:
Dark adaptation recovery time is a sensitive marker of AMD progression in intermediate AMD, largely owing to drusen volume providing a transport barrier that slows the transfer of nutrients between the choroid and photoreceptors2. Consequently, dark adaptation may provide an early indication of response vs. nonresponse, aiding case-by-case decisions on continuation of treatment when patients experience adverse side effects (e.g., elevated CPK or liver enzymes) or when atorvastatin provides insufficient lipid control in patients also at high-risk for cardiovascular disease (and switching to an alternative statin might be desirable).

ELIGIBILITY:
Inclusion Criteria:

* All subjects with intermediate AMD diagnosis in one or both eyes will be considered, regardless the severity stage and subtype of disease in the other eye.

High-risk iAMD (numerous large, confluent drusen covering ≥ 0.5 disk area, with or without pigmentary changes but having no evidence of GA or CNV) in the study eye

Subjects can have either:

(i) Bilateral high-risk iAMD, or (ii) High-risk iAMD in one eye with GA and/or CNV in the fellow eye.

Exclusion Criteria:

* Patient previously taking high dose Atorvastatin 80 mg
* Patients previously taking other statins than high dose atorvastatin, in whom primary care provider (PCP) feels cannot be safely moved to high dose atorvastatin or those in which high dose atorvastatin is deemed contraindicated by PCP
* Patients with known adverse reaction to statins
* Patients with severe renal disease or multiple comorbidities
* Age >85 years
* Pregnancy
* Patients with concomitant use of cyclosporine
* Active uveitis;
* Ocular infection;
* Any retinopathy other than AMD;
* Media opacities;
* Refractive error equal or superior to 6 diopters (spherical equivalent);
* Any previous retina surgery;
* Other ocular surgery or intra-ocular procedure in the study eye (injection other than anti angiogenic injection, laser) within the 90 days prior to enrollment

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Dark Adaptation recovery time measured by change in Rod Intercept time (RIT) | 18 Months
  Determine weather improvement in dark adaptation recovery time or rod intercept time (RIT) can be used as an early indicator of positive response to high dose statin therapy for intermediate AMD patients
Change in drusen volume measured by Spectral Domain OCT | 18 months
  To measure and quantify improvement or positive response to high dose statin therapy in patients with intermediate AMD using drusen volume measured by SDOCT
To correlate visual functions of dark adaption with change in drusen volume | 18 months
  Patient will have Dark Adaptation testing performed to check change in vision function with changes in drusen volume.

SECONDARY OUTCOMES:
To correlate Best Corrected Visual Acuity and retinal structural evaluation of study patients | 18 months
  Patient will have Best Corrected visual acuity, testing performed to check changes in vision function
To correlate change in contrast sensitivity and retinal structural evaluation of study patients | 18 months
  Patient will have quantitative contrast sensitivity function testing performed to check change in vision function with changes in drusen volume.
To correlate change in microperimetry visual functional and retinal structural evaluation of study patients | 18 months
  Patient will have microperimetry function testing performed to check change in this vision function with changes in drusen volume

CONTACTS AND LOCATIONS:
Overall Officials: John B Miller, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary, Harvard Medical School
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vavvas DG, Daniels AB, Kapsala ZG, Goldfarb JW, Ganotakis E, Loewenstein JI, Young LH, Gragoudas ES, Eliott D, Kim IK, Tsilimbaris MK, Miller JW. Regression of Some High-risk Features of Age-related Macular Degeneration (AMD) in Patients Receiving Intensive Statin Treatment. EBioMedicine. 2016 Feb 4;5:198-203. doi: 10.1016/j.ebiom.2016.01.033. eCollection 2016 Mar. PMID 27077128